CLINICAL TRIAL: NCT03939117
Title: Assessing the Feasibility and Safety of Using Intraoperative Ultrasound in Ileocolic Crohn's Disease - The IUSS Crohn's Feasibility Study
Brief Title: The IUSS Crohn's Study: A Feasibility Study
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2018/44
Record Dates: First submitted 2019-03-26; First posted 2019-05-06 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate if an intraoperative protocol for Ultrasound scan (USS) is feasible and safe in patients undergoing elective surgery for ileocolic CD. The results of this study could guide the development of a larger randomised trial.

DETAILED DESCRIPTION:
To date the intraoperative clinical assessment of location and extent of ileocolic CD has been left at the discretion of the operating surgeon guided by a mixture of experience, tactile feedback, macroscopic appearance and results of preoperative imaging, with significant intra and inter surgeon variability, potentially resulting in long segments of small bowel being removed unnecessarily, which is a significant concern in patients at risk of several abdominal surgeries and of developing "short bowel syndrome". At surgery, the operating surgeon also evaluates the full length of the small bowel to locate and assess further areas of CD: a process called "disease mapping". This process is not only important to intervene simultaneously on other CD segments causing complications, but also to provide the IBD MDT team with a full evaluation of the extent and severity of CD in that particular patient, in order to guide the tailored postoperative maintenance treatment.

A standardised approach to intraoperative evaluation of extent and location of CD is desirable, based on reliable and reproducible techniques, minimising the risk of surgical recurrence, optimising the decision making on maintenance treatment and follow-up, protecting patients from unnecessary extended small bowel resections and risk of short bowel syndrome.

The study objectives are To evaluate the feasibility of using intraoperative USS in patients with CD of the small bowel, and to describe the steps of the procedure.

To assess safety of the intraoperative USS procedure during surgery. To evaluate the feasibility of study delivery, i.e. recruitment of study participants and retention at follow-up visits.

To record surgical and patient outcomes up to 6 weeks To evaluate the direct and indirect costs of a standardised intraoperative USS protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over
2. American society of Anaesthesiologists (ASA) grade I, II or III
3. Undergoing elective surgery to remove part of the terminal ileum which is affected by CD.
4. . Indication for surgery agreed at IBD MDT meeting
5. Able to give written informed consent

Exclusion Criteria:

1. Undergoing emergency surgery
2. Previous abdominal surgery for CD
3. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is adults (18+ years) undergoing elective surgery (i.e. planned operation) for CD affecting the small bowel.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Number of intraoperative USS assessments completed. | Day of surgery
  Recording the number of intraoperative surgery completed
Number of adverse events reported during surgery. | Day of surgery
  Recording the number of adverse events reported during the surgey
To record the incidence of crohn's disease identified at macroscopic intraoperative assessment of the small bowel by the surgeon, and the intraoperative USS assessment of the small bowel. | Day of surgery
  recording the incidence of crohn's disease identified following assessment of the small bowel by the surgeon macroscopcially
To record the length of areas affected by crohn's disease identified at macroscopic intraoperative assessment of the small bowel by the surgeon | Day of surgery
  Measurement in centimeters of the length of bowel affected by crohn's disease as identified by the surgeon macroscopically
To compare the incidence of crohn's disease indentified macroscopically by the surgeon with the intraoperative ultrasound assessment | Day of surgery
  compare the incidence of crohn's disease identified by the surgeon with the incidence of crohn's disease identified by the intraoperative ultrasound assessment
To compare the length of crohn's disease identified marcoscopically by the surgeon with the intraoperative ultrasound assessment | Day of surgery
  compare the length of crohn's disease in centimetres identified by the surgeon with the incidence of crohn's disease identified by the intraoperative ultrasound assessment
To evaluate the feasibility of study delivery, i.e. recruitment of study participants and retention at follow-up visits. | 6 week follow up
  Feasibility of data collection required for a future trial measured by number of eligible participants, the proportion of patients consenting for the study, the proportion of recruited participants with all the required baseline and follow-up assessments completed, proportion of withdrawals from follow-up data collection, reasons for withdrawal and number of losses to follow-up.
To record surgical and patient outcomes up to 6 weeks | 30 day morbidity
  Operating time (Kaplan-Meier analysis), intra- and post-operative complication rates, 30 day morbidity and mortality rate
To evaluate the direct and indirect costs of a standardised intraoperative USS protocol. | 1 year
  Annotation of key steps for performance of small bowel intraoperative USS in patients with CD.

CONTACTS AND LOCATIONS:
Overall Officials: Valerio Celentano, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom